CLINICAL TRIAL: NCT03375697
Title: A 2-Part Randomized, Placebo-Controlled, Double-Blind, Single and Multiple Ascending Dose Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-63733657 in Healthy Subjects and Subjects With Alzheimer's Disease
Brief Title: A Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-63733657 in Healthy Subjects and Subjects With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR108392; 63733657EDI1001 (Other: Janssen Research & Development, LLC); 2017-003852-21 (EudraCT Number)
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD (Part 1): Healthy Subjects (Experimental): In Part 1, single ascending intravenous (IV) doses of JNJ-63733657 or placebo will be administered to sequential cohorts (Cohorts 1 to 5) of healthy subjects on Day 1. The progression to the next (higher) dose level is dependent on acceptable safety and tolerability profile of JNJ-63733657 obtained after dose administration of the current dose level. Here, SAD indicates single ascending dose.
  Interventions: Drug: JNJ-63733657; Drug: Placebo
- MAD (Part 2): Subjects With Alzheimer's Disease (AD) (Experimental): In Part 2, multiple ascending IV doses of JNJ-63733657 or placebo will be evaluated at three dose levels in sequential cohorts in subjects with prodromal or mild AD; 3 doses will be administered over a period of 8 weeks (Day 1, Day 29, Day 57). The starting dose will be decided based on the data from Part 1. Escalations will be done based on safety and tolerability similar to Part 1. Doses will not exceed those tested in Part 1. Here, MAD indicates multiple ascending dose.
  Interventions: Drug: JNJ-63733657; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-63733657 — Subjects will receive single (Part 1) or multiple (Part 2) ascending dose levels of JNJ-63733657 intravenously.
Drug: Placebo — Subjects will receive matching placebo intravenously.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of JNJ-63733657 following single ascending intravenous (IV) dose administration in healthy subjects (Part 1) and multiple ascending IV dose administrations in subjects with prodromal or mild Alzheimer's disease (AD) (Part 2).

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

* Body mass index (BMI) between 18 and 35 kilogram per meter square (kg/m^2), inclusive (BMI = weight/height^2) and body weight greater than 40 kilogram (kg) but less than 110 kg at screening
* Women must not be of childbearing potential

Specific Inclusion Criteria Part 2:

Each potential subject enrolled in Part 2 must satisfy all of the following specific criteria in addition to the general criteria to be enrolled in the study:

* Clinical Dementia Rating Scale (CDR) global rating score of 0.5 or 1.0 at screening
* Must have a reliable informant (example, relative, partner, friend)
* Must have cerebrospinal fluid (CSF) finding consistent with Alzheimer's disease (AD) pathology

Exclusion Criteria:

General Exclusion Criteria

Any potential subject who meets any of the following criteria will be excluded from participating in the study:

* History of or current liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic (including but not limited to neurodegenerative disease (excluding AD for Part 2) [example, Parkinson's disease], seizure disorders, transient ischemic attacks, etc.), hematologic (including coagulation disorders), rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness that the Investigator considers should exclude the subject
* Relevant history of or current neurological disease (other than prodromal AD or mild AD for Part 2), which in the opinion of the investigator may make interpretation of possible new neurological signs or symptoms difficult
* History of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening (per screening evaluations)
* History of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-Hepatitis C virus [HCV]) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening (per screening evaluations)

Specific Exclusion Criteria Part 1 - Mini-Mental State Examination (MMSE) score less than or equal to (<=) 27 at screening

Specific Exclusion Criteria Part 2

- Evidence of brain disease, other than AD, that could explain the cognitive deficit (including, but not limited to, vascular encephalopathy or strokes, as imaged by cerebral Magnetic resonance imaging (MRI)

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Single Ascending Dose (SAD) (Part 1): Number of Subjects With Adverse Events as a Measure of Safety and Tolerability of JNJ-63733657 | Up to Day 106
  An adverse event is any untoward medical event that occurs in a subject administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Multiple Ascending Dose (MAD) (Part 2): Number of Subjects With Adverse Events as a Measure of Safety and Tolerability of JNJ-63733657 | Up to Day 162
  An adverse event is any untoward medical event that occurs in a subject administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
SAD (Part 1) and MAD (Part 2): Maximum Observed Serum Concentration (Cmax) of JNJ-63733657 | Up to Day 106 (SAD) and up to Day 162 (MAD)
  The Cmax is the maximum observed serum concentration of drug JNJ-63733657.
SAD (Part 1) and MAD (Part 2): Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-63733657 | Up to Day 106 (SAD) and up to Day 162 (MAD)
  Tmax is defined as time to reach the maximum observed serum JNJ-63733657 concentration.
SAD (Part 1) and MAD (Part 2): Area Under the Serum Concentration-time Curve From Time Zero to Time of the Last Observed Quantifiable Concentration (AUC [0-Last]) of JNJ-63733657 | Up to Day 106 (SAD) and up to Day 162 (MAD)
  AUC (0-last) is defined as area under the serum JNJ-63733657 concentration-time curve from time 0 to time of the last observed quantifiable concentration.
SAD (Part 1) and MAD (Part 2): Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-63733657 | Up to Day 106 (SAD) and up to Day 162 (MAD)
  AUC (0-infinity) is defined as area under the serum JNJ-63733657 concentration-time curve from time 0 to infinite time.
MAD (Part 2): Area Under the Serum JNJ-63733657 Concentration-time Curve During a Dosing Interval (t) (AUC tau) | Up to Day 85 (MAD)
  AUC tau is defined as area under the serum JNJ-63733657 concentration-time curve during a dosing interval (tau).
MAD (Part 2): Accumulation Ratio (R) | Up to Day 162 (MAD)
  R is obtained by dividing AUC of JNJ-63733657 at two different time points.
SAD (Part 1) and MAD (Part 2): Total Systemic Clearance (CL) of JNJ-63733657 | Up to Day 106 (SAD) and up to Day 162 (MAD)
  CL is a quantitative measure of the rate at which JNJ-63733657 is removed from the body. The total systemic clearance after intravenous dose is estimated by dividing the total administered dose by the plasma Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]).
SAD (Part 1) and MAD (Part 2): Volume of Distribution at Steady-State (Vss) of JNJ-63733657 | Up to Day 106 (SAD) and up to Day 162 (MAD)
  Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state Vss is the apparent volume of distribution at steady-state which is estimated by (D/AUC[0-infinity])*(AUMC[0-infinity])/AUC[0-infinity]) where D is the dose of study drug, AUMC(0-infinity) is the area under the first moment curve extrapolated to infinity and AUC(0-infinity) is the area under the serum concentration-time curve from time zero to infinite time.
SAD (Part 1) and MAD (Part 2): Terminal Half-Life(t[1/2]) of JNJ-63733657 | Up to Day 106 (SAD) and up to Day 162 (MAD)
  t(1/2) is associated with the terminal slope (lambda [z]) of the semi-logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
SAD (Part 1) and MAD (Part 2): JNJ-63733657 Concentration in Cerebrospinal Fluid (CSF) | Up to Day 57 (SAD) and up to Day 148 (MAD)
  CSF concentration assessment will be done to characterize the pharmacokinetics (PK) to estimate CSF concentration of JNJ-63733657.
SAD (Part 1) and MAD (Part 2): Number of Subjects With Anti-JNJ-6373365 Antibodies as a Measure of Immunogenicity | Up to Day 106 (SAD) and up to Day 162 (MAD)
  Number of subjects with Anti-JNJ-63733657 antibodies will be evaluated in serum samples and potential CSF samples.
SAD (Part 1) and MAD (Part 2): Percent Change From Baseline in Total, Free, and Bound tau Biomarker Fragments in CSF | Up to Day 106 (SAD) and up to Day 162 (MAD)
  Percent change from baseline in total, free, and bound tau (phosphorylation site) biomarker fragments in CSF will be evaluated to assess the effect of JNJ-63733657.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (7):
- Clinical Pharmacology Unit, Merksem, Belgium
- Germany (3):
  - Klinik für Neurodegenerative Erkrankungen und Gerontopsychiatrie, Bonn
  - CTC North GmbH & Co. KG, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg / Saar
- Centre for Human Drug Research, Leiden, Netherlands
- Spain (2):
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. I Politecni La Fe, Valencia